CLINICAL TRIAL: NCT00530504
Title: Carotid Revascularization With ev3 Arterial Technology Evolution Post Approval Study
Acronym: CREATE PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-2611
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Carotid Artery Disease
Keywords: Carotid Artery Disease; Embolic Protection
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Experimental): Device
  Interventions: Device: PROTÉGÉ™ GPS™ and PROTÉGÉ™ RX Carotid Stent Systems and SpiderFX™ Embolic Protection Device

INTERVENTIONS:
Device: PROTÉGÉ™ GPS™ and PROTÉGÉ™ RX Carotid Stent Systems and SpiderFX™ Embolic Protection Device — Carotid artery stenting with distal embolic protection.

SUMMARY:
The purposes of this study are:

1. To provide additional safety and effectiveness information on the commercial use of Protégé™ GPS™ and Protégé™ RX Carotid Stent Systems and the SpiderFX™ Embolic Protection Device.
2. To evaluate rare and unanticipated adverse events.
3. To evaluate the physician level of experience with carotid artery stenting procedures with adverse event rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Informed consent
* Intent to use the PROTÉGÉ™ GPS™ and PROTÉGÉ™ RX and SpiderFX™ to treat carotid artery disease per Instructions for Use
* Meet Instruction for Use (IFU)/ Centers for Medicare & Medicaid Services (CMS)defined anatomical or clinical high risk criteria

Exclusion Criteria:

* Subjects with contraindications as outlined in the Instructions for Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2007-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ansel, MD, Principal Investigator — MidWest Cardiology Research Foundation; Robert Safian, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Stony Brook University Hospital, Stony Brook, New York
  - Wellmont Medical Center, Kingsport, Tennessee

REFERENCES:
- See also: Click here for information on ev3 Endovascular Inc. — http://www.ev3.net

RESULTS

PARTICIPANT FLOW:
Groups:
- Stent and Protection Device: PROTÉGÉ™ GPS™ and PROTÉGÉ™ RX Carotid Stent Systems and SpiderFX™ Embolic Protection Device: Carotid artery stenting with distal embolic protection.
Period: Overall Study
Arm/Group | Stent and Protection Device
Started | 1500
Completed | 1348
Not Completed | 152
Not completed — Death | 54
Not completed — Lost to Follow-up | 26
Not completed — Withdrawal by Subject | 39
Not completed — Exited study due to other reasons | 33

BASELINE CHARACTERISTICS:
Groups:
- Intervention: PROTÉGÉ™ GPS™ and PROTÉGÉ™ RX Carotid Stent Systems and SpiderFX™ Embolic Protection Device: Carotid artery stenting with distal embolic protection.
Arm/Group | Intervention
Number analyzed (Participants) | 1500
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 577
  Male | 923

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Death, Ipsilateral CVA, Procedure-related CVA, or Myocardial Infarction (MI) at 30 Days Post-procedure.
Description: Combined incidence of Major Adverse Cardiac and Cerebrovascular Events (MACCE) defined as myocardial infarction (MI), ipsilateral cerebrovascular accident (CVA), procedure-related contralateral CVA, or death, within 30 days of implantation.
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 1500
participants | 99

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 553/1500
Other Adverse Events (participants affected / at risk) | 258/1500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1500)
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 33 (34)
Cardiac disorder (Cardiac disorders) | 98 (117)
Ear And Labyrinth Disorders (Ear and labyrinth disorders) | 2 (2)
Eye disorder (Eye disorders) | 8 (8)
Gastrointestinal disorders (Gastrointestinal disorders) | 35 (42)
General Disorders And Administrative Site Conditions (General disorders) | 71 (76)
Hepatobiliary disorders (Hepatobiliary disorders) | 4 (5)
Immune System Disorders (Immune system disorders) | 2 (2)
Infections And Infestations (Infections and infestations) | 46 (51)
Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 19 (20)
Investigations (Investigations) | 15 (16)
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 10 (10)
Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 12 (12)
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Nervous System Disorders (Nervous system disorders) | 142 (150)
Psychiatric Disorders (Psychiatric disorders) | 11 (11)
Renal And Urinary Disorders (Renal and urinary disorders) | 26 (28)
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 30 (33)
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 3 (3)
Surgical And Medical Procedures (Surgical and medical procedures) | 29 (29)
Vascular Disorders (Vascular disorders) | 268 (284)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1500)
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 13 (13)
Cardiac disorders (Cardiac disorders) | 24 (24)
Ear And Labyrinth Disorders (Ear and labyrinth disorders) | 3 (3)
Eye Disorders (Eye disorders) | 17 (17)
Gastrointestinal Disorders (Gastrointestinal disorders) | 25 (27)
General Disorders And Administrative Site Conditions (General disorders) | 40 (41)
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1)
Immune System Disorders (Immune system disorders) | 2 (2)
Infections And Infestations (Infections and infestations) | 39 (47)
Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 12 (12)
Investigations (Investigations) | 16 (17)
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 7 (8)
Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 29 (35)
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Nervous System Disorders (Nervous system disorders) | 44 (46)
Psychiatric Disorders (Psychiatric disorders) | 7 (7)
Renal And Urinary Disorders (Renal and urinary disorders) | 19 (20)
Reproductive System And Breast Disoders (Reproductive system and breast disorders) | 1 (1)
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 24 (27)
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 10 (11)
Surgical And Medical Procedures (Surgical and medical procedures) | 10 (14)
Vascular Disorders (Vascular disorders) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results without permission of the sponsor.